CLINICAL TRIAL: NCT01878162
Title: Effectiveness of an Exercise-based Work Injury Prevention Program in Law Enforcement Officials
Brief Title: Work Injury Prevention in Law Enforcement Officials
Status: Suspended | Phase: Not Applicable | Type: Interventional
Sponsor: University of the Pacific (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: UPacific_Davenport1
Record Dates: First submitted 2012-08-03; First posted 2013-06-14 (Estimated); Last update posted 2015-07-02 (Estimated); Status verified 2015-07

CONDITIONS: Exercise
Keywords: Prevention; Wellness; Occupation; Work; Law Enforcement; Exercise
MeSH Terms: conditions — Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Exercise (Experimental): Exercise will occur 3 times weekly for 6 months in 20-minute exercise sessions. Sessions will take place independently. Follow-up and progression of the home program will be completed in person or by video teleconferencing at regular intervals throughout the intervention phase.
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise

SUMMARY:
Law enforcement officials (LEOs) demonstrate an elevated risk for occupational injury. The effectiveness of exercise-based work injury prevention programs (WIPPs) to reduce the risk and costs associated with occupational injury has yet to be tested rigorously in LEOs. The accuracy of existing field tests of physical functioning to predict occupational injuries and related expenses remains unclear. The objectives of this study are to: (i) determine the effect of an exercise-based WIPP on occupational wellness and productivity in a cohort of LEOs, and (ii) to determine the accuracy of 2 common field assessments of physical function to predict lost work productivity and related expenses in a cohort of LEOs.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 60 years
* Working full duty as a law enforcement official

Exclusion Criteria:

* Current history of pathology or symptoms that preclude exercise
* Medical or rehabilitative treatment for a work-related injury within the past year prior to enrollment in this study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 108 (Estimated)
Dates: Start 2012-08; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Number of Work Injury Claims During the Study Period | One time, at one year following enrollment into the study
Medical Expenditures Related to Work Injury Claims During the Study Period | One time, at one year following enrollment into the study
Number of Missed Work Days Due to Illness or Injury | One time, at one year following enrollment into the study
Work Productivity and Activity Impairment Questionnaire - General Health Subscale | Weekly, up to one year following enrollment into the study
  The Work Productivity and Activity Impairment (WPAI) Questionnaire was developed to measure the personal and economic effects of lost workplace productivity in the context of clinical trials. In this study, the WPAI-General Health (GH) version will be used in order to assess lost productivity and wellness during the study period. The WPAI-GH is a 6-item scale that solicits the number of hours missed from work and level of functional impairment perceived at work during the previous week. Four scores are calculated from the WPAI-GH, including percentage of work time missed due to health, percentage impairment while working due to health, percentage activity impairment due to health, an overall percentage work impairment. Time series data will be collected to observe trends over time that may relate to independent variables in this study, as well as to examine for previously unknown and uncontrolled variation (ie, seasonal variability).

SECONDARY OUTCOMES:
Functional Movement Screen | One time, at 3 months following enrollment into the study
  The purpose of the Functional Movement Screen (FMS) is to provide the clinician with a rapid triage for potentially problematic regions that can contribute to symptoms, disablement, or injury. As a triage tool, FMS is used to determine regions that require additional clinical investigation. The FMS is a battery of 7 tests that are intended as an integrated assessment for limitations in range of motion, weakness, and incoordination. FMS tests consider spine, upper extremity, and lower extremity movements in the context of their respective regional kinetic chain. Component tests of the FMS involve rating of performance by a standardized examiner on a 3-point scale, and specific criteria exist for each rating. A composite score for the FMS may be calculated by summing the item scores.
Star Balance Excursion Test | One time, at 3 months following enrollment into the study
  The Star Excursion Balance Test is a clinical test of dynamic balance. Subjects will assume unilateral stance in the center of a grid marked circumferentially in 45-degree increments. After a learning trial consisting of 6 repetitions in each of the 8 test directions, subjects will complete 3 repetitions of single limb squat reach. The evaluating therapist will record the distance achieved between the stance toe and heel of the reaching extremity in each of 3 repetitions in each direction.

CONTACTS AND LOCATIONS:
Overall Officials: Todd E Davenport, PT, DPT, OCS, Principal Investigator — University of the Pacific
Locations (5):
- United States (5):
  - Butte Premier Physical Therapy, Chico, California
  - Physical Edge, Davis, California
  - PUMP Institute, Lodi, California
  - Lodi Physical Therapy, Lodi, California
  - University of the Pacific, Stockton, California